CLINICAL TRIAL: NCT01234805
Title: Yoga and Brain Cancer: A Feasibility Study
Brief Title: Yoga Therapy in Treating Patients With Malignant Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00015038; NCI-2010-02044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98410 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Meningioma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Choroid Plexus Tumor; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade II Meningioma; Adult Medulloblastoma; Adult Meningeal Hemangiopericytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Papillary Meningioma; Adult Pineal Gland Astrocytoma; Adult Pineoblastoma; Adult Pineocytoma; Adult Supratentorial Primitive Neuroectodermal Tumor (PNET); Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Choroid Plexus Neoplasms; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Glioma; Pinealoma; Brain Neoplasms | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (yoga therapy) (Experimental): Patients participate in yoga classes comprising postures, deep relaxation, breathing practices, and meditation twice weekly for 75 minutes during weeks 1-6. Patients then practice yoga at home twice weekly for 45 minutes during weeks 7-12.
  Interventions: Procedure: yoga therapy; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: yoga therapy — Participates in yoga classes and yoga at home
  Other Names: yoga
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This clinical trial studies yoga therapy in treating patients with malignant brain tumors. Yoga therapy may improve the quality of life of patients with brain tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the participation rate, accrual, adherence, and retention to a yoga trial in patients with malignant brain tumors.

SECONDARY OBJECTIVES:

I. To obtain estimates of the variability of self-reported fatigue, distress (i.e., depression, anxiety), sleep disturbance, cognitive function, and health-related quality of life from baseline to the end of the intervention at 6 (post-onsite intervention) and 12 weeks (post-full intervention).

II. To obtain preliminary estimates of the efficacy of a yoga intervention in patients with malignant brain tumors on the outcomes of fatigue, distress, and cognitive function.

III. To standardize the cancer-specific yoga protocol for use with brain tumor patients.

OUTLINE:

Patients participate in yoga classes comprising postures, deep relaxation, breathing practices, and meditation twice weekly for 75 minutes during weeks 1-6. Patients then practice yoga at home twice weekly for 45 minutes during weeks 7-12.

After completion of study treatment, patients are followed up periodically for 4-5 months.

ELIGIBILITY:
Inclusion Criteria:

Signed protocol specific informed consent Are diagnosed with a Malignant Brain Tumor (Grades II-IV) Able to start the on-site yoga intervention within 1 week of first radiation treatment Are physically able to attend the intervention classes (Eastern Cooperative Oncology Group [ECOG] performance status rating 0-2) Able to understand written and spoken English Have no medical contraindications reported by the attending physician

Exclusion Criteria:

Have practiced yoga on a regular basis (at least once a week) within the past 4 weeks to recruit participants who are not already regularly practicing yoga; given that the benefits of yoga are likely more immediate than long-term, however, we will enroll participants who have previously had a yoga practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Estimate the participation rate, accrual, adherence, and retention to a yoga trial in patients with malignant brain tumors | Up to 12 weeks
  Track barriers to recruitment. Participation rate calculated as proportion of eligible patients who agree to participate. Study retention estimated as proportion of participating patients who complete questionnaires at Week 6. Further retention data obtained by tracking # of dropouts, when dropout occurs, & reasons for dropout. Intervention adherence estimated as mean % of yoga classes attended. Summary statistics for patient characteristics, participation rates, adherence & retention. 95% confidence intervals calculated for each feasibility measure.

SECONDARY OUTCOMES:
Self-reported fatigue | Up to 12 weeks
Depressive symptoms | Up to 12 weeks
Distress | Up to 12 weeks
Health-related quality of life | Up to 12 weeks
Preliminary estimates of the efficacy of a yoga intervention in patients with malignant brain tumors on the outcomes of fatigue, distress, and cognitive function | Up to 12 weeks
Standardize the cancer-specific yoga protocol for use with brain tumor patients | At the end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States